CLINICAL TRIAL: NCT05447182
Title: People-Powered Medicine (PPM): Rheumatoid Arthritis Non-responders to Biologic Therapies (RANT)
Acronym: PPM:RANT
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Katherine P Liao, Associate Professor of Medicine and Biomedical Informatics, Brigham and Women's Hospital
Other Study IDs: IRB20-1219
Record Dates: First submitted 2021-08-05; First posted 2022-07-07 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Treatment non-response; Tumor necrosis factor inhibitor (TNFi); Rheumatoid Arthritis; Disease modifying anti-rheumatic therapy; Biologic therapy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One-time blood draw to measure proteomics and conduct whole genome sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are interested in enrolling patients with rheumatoid arthritis (RA) who had a difficult time getting their disease under control even after trying multiple RA therapies. The investigators believe that there may be common patterns in the genes of this group of RA patients compared to those with more "textbook RA." Understanding genetic factors can help doctors to know in advance who may not respond to conventional therapies and start with treatments that work. Learning about underlying genes that influence treatment may help the investigators to identify new targets for therapy, to ultimately improve the lives of patients with RA and inflammatory arthritis.

DETAILED DESCRIPTION:
The investigators are looking for patients with rheumatoid arthritis (RA) with an inadequate response to tumor necrosis factor inhibitor (TNFi) and another biologic disease modifying anti-rheumatic drug (bDMARD) or small molecule approved for treating RA. The investigators are conducting this research to learn more about RA and the genetic patterns associated with patients whose RA cannot be well controlled with most RA treatments. Investigators anticipate that these patients will differ from "classic" RA patients in their biomarker and genetic composition and that they represent a mixed group of individuals who may be similar in ways that are not currently being measured.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* RA diagnosed by a rheumatologist
* Poor control of RA disease activity with tumor necrosis factor inhibitor (TNFi) and another biologic therapy or small molecule approved for RA

Exclusion Criteria:

* If the reason for failed TNFi therapy was due to a contraindication or adverse reaction
* Unable to provide blood sample

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Study Population: Patients diagnosed with rheumatoid arthritis (RA) that have failed TNFi therapy and another bDMARD or small molecule approved for RA.
  TNFi= adalimumab (Humira), certolizumab (Cimzia), etanercept (Enbrel), infliximab (Remicade), golimumab (Simponi)
  bDMARDs or small molecules for RA in addition to TNFi above: abatacept (Orencia), baricitinib (Olumiant), sarilumab (Kevzara), tocilizumab (Actemra), rituximab (Rituxan), tofacitinib (Xeljanz), upadacitinib (Rinvoq)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Whole genome sequencing | Through study completion, averaging 1 year
  Genomic data will be applied in an established bioinformatics pipeline to screen for uncommon variants and test association with exceptional treatment non-responders compared with TNFi responders.

SECONDARY OUTCOMES:
Subgroup analyses of treatment non-responders | 1 year
  Patients who eventually find a therapy that controls their RA. The investigators will use prospective questionnaire data to subgroup patients into those who eventually find a treatment that works vs those who do not.

OTHER OUTCOMES:
Other potential predictors of poor response to biologic therapies | Retrospective data up to 10 years prior to enrollment
  Electronic health data will be used to assess for common features of patients who have poor response to therapy compared to TNFi responders.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McDermott GC, Jeffway M, Seyok T, Zhang H, Myasoedova E, Davis JM 3rd, Giles J, Coblyn J, Helfgott S, Massarotti E, Sands R, Weinblatt ME, Johansson T, Schmajuk G, Michaud K, Perry C, Churchill S, Liao KP. Rationale and design of the rheumatoid arthritis non-responders to treatment (RANT) study: Use of a bioinformatics platform and "decentralized" clinical recruitment design. Contemp Clin Trials. 2025 Sep;156:108000. doi: 10.1016/j.cct.2025.108000. Epub 2025 Jul 14. PMID 40669748